CLINICAL TRIAL: NCT02740387
Title: A 1-Year, Phase 2, Open-Label Safety Study of OTO-104 Given at 3-Month Intervals by Intratympanic Injection in Subjects With Unilateral Meniere's Disease
Brief Title: Open Label Study of OTO-104 in Subjects With Meniere's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Negative Efficacy Results from the recently completed Phase 3 study 104-201506
Sponsor: Otonomy, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 104-201505
Record Dates: First submitted 2016-03-25; First posted 2016-04-15 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Meniere's Disease
MeSH Terms: conditions — Meniere Disease | interventions — Injection, Intratympanic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OTO-104 (Experimental): 12 mg dexamethasone
  Interventions: Drug: OTO-104

INTERVENTIONS:
Drug: OTO-104
  Other Names: Single intratympanic injection 12 mg OTO-104

SUMMARY:
This is a 1-year, multicenter, Phase 2, open-label safety study in subjects with unilateral Meniere's disease. Subjects will receive 1 intratympanic (IT) injection of 12 mg OTO-104 at 3-month intervals for a total of 4 injections total.

ELIGIBILITY:
Inclusion Criteria includes, but is not limited to:

* Subject has a diagnosis of definite unilateral Meniere's disease.
* Subject agrees to maintain their current standard of care treatments for Meniere's disease while on-study.

Exclusion Criteria includes, but is not limited to:

* Subject has an infection in the ear, sinuses, or upper respiratory system.
* Subject is pregnant or lactating.
* Subject has a history of immunodeficiency disease.
* Subject has active or recent (<1 month prior to screening) middle ear disease, including but not limited to: chronic otitis media, acute otitis media, middle ear effusions, middle ear atelectasis, or cholesteatoma.
* Subject has experienced an adverse reaction to intratympanic injection of steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of adverse events as a measure of safety and tolerability | Up to 1 Year

SECONDARY OUTCOMES:
Change in hearing from baseline as assessed by audiometry | Up to 1 Year
Changes in patient condition assessed by otoscopy | Up to 1 Year
Changes in patient condition assessed by tympanometry | Up to 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Kathie Bishop, PhD, Study Chair — Otonomy, Inc.
Locations (1):
- Call Otonomy call center for trial locations, London, Ontario, Canada